CLINICAL TRIAL: NCT00516659
Title: A Phase II, Double Blind, Randomized, Placebo-Controlled Study to Evaluate the Epidemiology of Natural Infection With Enterotoxigenic Escherichia Coli Occurring After Transcutaneous Immunization in a Field Setting
Brief Title: ETEC Logistics Trial (TREK)
Acronym: Trek
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: ELT206
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Diarrhea
Keywords: ETEC; Traveler's diarrhea; TCI; patch vaccine; diarrhea prevention; epidemiology ETEC; Escherichia coli
MeSH Terms: conditions — Diarrhea; Escherichia coli Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Group 1 subjects will receive two vaccinations via transcutaneous immunization (TCI), 14 to 21 days apart, with a patch containing 37.5µg LT
  Interventions: Biological: Heat-Labile Enterotoxin of Escherichia coli (LT)
- Group 2 (Placebo Comparator): Group 2 subjects will receive two vaccinations via transcutaneous immunization (TCI), 14 to 21 days apart, with a patch containing 0µg LT (placebo patch containing no LT)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Heat-Labile Enterotoxin of Escherichia coli (LT) — Subjects in Group 1 will receive two vaccinations of a patch containing 37.5µg LT 2 to 3 weeks apart.
  Arms: Group 1
Biological: Placebo — The placebo patch contains all of the components of the active patch, but with no LT included in the formulation.
  Arms: Group 2

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled field trial to evaluate the epidemiology of natural infection with ETEC occurring after transcutaneous immunization in a field setting.

DETAILED DESCRIPTION:
The primary objectives of the study are to evaluate the incidence of ETEC illness in a field setting and to compare the safety of LT delivered by TCI with placebo. The secondary objectives include, but are not limited to:

evaluate the stool frequency per episode of ETEC illness in placebo recipients, to evaluate the immunogenicity of LT delivered by TCI, to evaluate the incidence of IBS following travel to areas of ETEC endemnicity, and to evaluate the incidence of VPO in placebo and LT patch recipients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women 18-64 years of age inclusive at screening
* Signed Informed Consent form
* Planned travel to an area within 2 ½ hours traveling distance of Cuernavaca or Guadalajara, Mexico or Antigua, Guatemala (minimum stay of 7 days)
* If female who is not post-menopausal or surgically sterile, negative pregnancy test (within 24 hours prior to vaccination) and agreement to employ an effective form of birth control or practice abstinence through the end of the study.

Exclusion Criteria:

* Clinically significant abnormalities as determined by the Investigator/clinician during physical inspection
* Received investigational product from 30 days before date of first vaccination or during the entire study period
* Ever received LT, ETEC, or cholera vaccine
* History of traveler's diarrhea within the previous year
* Travel to a developing country within the last year
* Women who are pregnant or breastfeeding
* History of achlorhydria
* Evidence of immunosuppression, including concomitant immunosuppressive therapy; fever > 99.5°F (37.5°C) on day of vaccination
* Current problems with alcohol or substance abuse
* An employee of the study clinic
* Sensitivity or allergy to any of the vaccine components
* History of significant blood loss, blood product donation, or blood product recipient in the previous 60 days
* Planned use of Imodium or antibiotics for self treatment of diarrhea during the study period
* Visible tattoos or marks (tattoos/scars) at the vaccination areas that would prevent appropriate dermatologic monitoring of the vaccination sites; and
* Medical history of acute or chronic GI illness or major GI surgery.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Enterotoxigenic Escherichia coli (ETEC) illness defined as a diarrheal episode associated with an LT, LT/ST, or ST-positive ETEC strain isolated from a sample of a stool | during the diarrheal episode or within 48 hours after the last stool in the diarrheal episode.
Safety of heat-labile enterotoxin of Escherichia coli (LT) delivered by transcutaneous immunization (TCI) vs placebo | From vaccination 1 to completion of Day 180 follow-up, about a seven month time period

SECONDARY OUTCOMES:
Stool frequency per episode of ETEC illness in placebo recipients | Duration of stay in Mexico or Guatemala assessed up to four weeks
Immunogenicity of LT delivered by TCI | at least three weeks prior to arrival in country, arrival in Mexico or Guatemala, and 5 to 18 days after arrival
Incidence of irritable bowel syndrome following travel to areas of ETEC endemnicity. | Baseline through six months post return from Latin America. A period of about six months.
Incidence of vaccine preventable outcome in placebo and LT patch recipients. | Duration of each individual participant stay in Mexico or Guatemala ranging from 7 to 28 Days.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L. DuPont, MD, Principal Investigator — Center for Infectious Diseases, The University of Texas Health Science Center at Houston; Robin McKenzie, MD, Principal Investigator — Johns Hopkins University, Bloomberg School of Public Health; Rama Yerramsetti, Principal Investigator — Breco Research, Houston, TX; William P Jennings, Principal Investigator — Radiant Research, San Antonio, TX; Yu-Luen Hsu, Principal Investigator — West Coast Clinical Trials, Long Beach, CA; Christopher A Smith, Principal Investigator — Asthma & Allergy Associates, Ithaca, NY; Benno G Roesch, Principal Investigator — Advanced Biomedical Research, Hackensack, NJ; Jeffrey G Geohas, Principal Investigator — Radiant Research, Chicago, IL; Gilbert Podolsky, Principal Investigator — Jean Brown Research, Salt Lake City, UT; Thomas Lagen, Principal Investigator — Northwest Kinetics, Tacoma, WA; Roy M Fleischmann, Principal Investigator — Radiant Research, Dallas, TX; Douglas R Schumacher, Principal Investigator — Radiant Research, Columbus, OH; Norman M Lunde, Principal Investigator — Twin Cities Clinical Research, Minneapolis, MN; Francisco G Sandoval, Principal Investigator — Universidad Autonoma De Guadalajara, Mexico; Juan Hector M Romero, Principal Investigator — Universidad Autonoma Guadalajara, Mexico; Jaime B Gerson, Principal Investigator — University of Texas, Cuernavaca, Mexico; Edwin Asturias, Principal Investigator — Universidad del Valle de Guatemala (Antigua); Roberto Garcia, Principal Investigator — AmeriMed Puerto Vallarta, Mexico; Martha V Serrato, Principal Investigator — Hospital Americano, Cancun, Mexico; Robert Maxwell, Principal Investigator — Private Clinic, San Miguel de Allende, Mexico
Locations (19):
- United States (13):
  - West Coast Clinical Trials, Long Beach, California
  - Radiant Research, Chicago, Illinois
  - Johns Hopkins University, Bloomberg School of Public Health, Baltimore, Maryland
  - Twin Cities Clinical Research, Minneapolis, Minnesota
  - Advanced Biomedical Research, Hackensack, New Jersey
  - Asthma Allergy & Associates, Ithica, New York
  - Radiant Research, Columbus, Ohio
  - Radiant Research, Dallas, Texas
  - Breco Research, Houston, Texas
  - Center for Infectious Diseases, The University of Texas Health Science Center at Houston, Houston, Texas
  - Radiant Research, San Antonio, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - Northwest Kinetics, Tacoma, Washington
- Private Clinic Antigua, Antigua Guatemala, Guatemala
- Mexico (5):
  - Private Clinic San Miguel, San Miguel de Allende, Guanajuata
  - Private Clinic Guadalajara, Guadalajara, Jalisco
  - AmeriMed Hospital, Puerto Vallarta, Marina Vallarta
  - Private Clinic Cuernavaca, Cuernavaca, Morelos
  - Hospital Americano, Cancún, Quintana Roo

REFERENCES:
- [Derived] Frech SA, Dupont HL, Bourgeois AL, McKenzie R, Belkind-Gerson J, Figueroa JF, Okhuysen PC, Guerrero NH, Martinez-Sandoval FG, Melendez-Romero JH, Jiang ZD, Asturias EJ, Halpern J, Torres OR, Hoffman AS, Villar CP, Kassem RN, Flyer DC, Andersen BH, Kazempour K, Breisch SA, Glenn GM. Use of a patch containing heat-labile toxin from Escherichia coli against travellers' diarrhoea: a phase II, randomised, double-blind, placebo-controlled field trial. Lancet. 2008 Jun 14;371(9629):2019-25. doi: 10.1016/S0140-6736(08)60839-9. PMID 18554712
- See also: Related Info — http://www.trekstudy.com